CLINICAL TRIAL: NCT02949284
Title: Randomized Three-Arm Trial to Evaluate the Effect of Neoadjuvant Apalutamide Alone or in Combination With Abiraterone Acetate and GnRH Agonist on Enhancing Surgical Outcome of Nerve-Sparing Radical Prostatectomy in Men With High-Risk Prostate Cancer
Brief Title: Androgen Receptor Antagonist ARN-509 With or Without Abiraterone Acetate, Gonadotropin-Releasing Hormone Analog, and Prednisone in Treating Patients With High-Risk Prostate Cancer Undergoing Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Saum Ghodoussipour, Professor of Surgery, RWJMS, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro20160000563; NCI-2016-01496 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20160000563; 081603 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2016-10-21; First posted 2016-10-31 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Stage II Prostate Adenocarcinoma; Stage III Prostate Adenocarcinoma
MeSH Terms: interventions — Abiraterone Acetate; apalutamide; Gonadotropin-Releasing Hormone; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (androgen receptor ARN-509, radical prostatectomy) (Experimental): Patients receive androgen receptor antagonist ARN-509 PO daily for 3 months. Patients then undergo radical prostatectomy.
  Interventions: Drug: Androgen Receptor Antagonist ARN-509; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Radical Prostatectomy
- Arm II (ARN-509, abiraterone acetate, GnRH, prednisone, RP) (Active Comparator): Patients receive GnRH agonist SC on day 1, androgen receptor antagonist ARN-509 PO daily PO for 4 times, abiraterone acetate PO daily for 4 times, and prednisone PO daily for 3 months. Patients then undergo radical prostatectomy.
  Interventions: Drug: Abiraterone Acetate; Drug: Androgen Receptor Antagonist ARN-509; Biological: Gonadotropin-releasing Hormone Analog; Drug: Prednisone; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Radical Prostatectomy
- Arm III (radical prostatectomy) (Active Comparator): Patients undergo radical prostatectomy.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Zytiga
  Arms: Arm II (ARN-509, abiraterone acetate, GnRH, prednisone, RP)
Drug: Androgen Receptor Antagonist ARN-509 — Given PO
  Other Names: ARN-509
  Arms: Arm I (androgen receptor ARN-509, radical prostatectomy); Arm II (ARN-509, abiraterone acetate, GnRH, prednisone, RP)
Biological: Gonadotropin-releasing Hormone Analog — Given SC
  Other Names: GnRH Agonist; GnRH Analog; Gonadotropin-Releasing Hormone Agonist; Gonadotropin-Releasing Hormone Analogue; LH-RH agonist; LH-RH Analogs; LHRH Agonist; luteinizing hormone-releasing hormone agonist; Luteinizing Hormone-Releasing Hormone Analog
  Arms: Arm II (ARN-509, abiraterone acetate, GnRH, prednisone, RP)
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
  Arms: Arm II (ARN-509, abiraterone acetate, GnRH, prednisone, RP)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Radical Prostatectomy — Undergo radical prostatectomy
  Other Names: Prostatovesiculectomy

SUMMARY:
This randomized phase II trial studies how well androgen receptor antagonist ARN-509 works with or without abiraterone acetate, gonadotropin-releasing hormone agonist, and prednisone in treating patients with high-risk prostate cancer undergoing surgery. Androgen can cause the growth of prostate cancer cells. Hormone therapy using androgen receptor antagonist ARN-509, abiraterone acetate, and gonadotropin-releasing hormone analog (GnRH agonist) may fight prostate cancer by lowering the levels of androgen the body makes. Prednisone may either kill the tumor cells or stop them from dividing. Giving androgen receptor agonist ARN-509 with or without abiraterone acetate, GnRH agonist and prednisone may work better in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of neoadjuvant androgen receptor antagonist ARN-509 (apalutamide) with or without abiraterone acetate, GnRH agonist, and prednisone on the feasibility of performing nerve-sparing radical prostatectomy (RP) in men with high-risk prostate cancer (PCa).

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive androgen receptor antagonist ARN-509 orally (PO) daily for 3 months. Patients then undergo radical prostatectomy.

ARM II: Patients receive GnRH agonist subcutaneously (SC) on day 1, androgen receptor antagonist ARN-509 PO daily PO for 4 times, abiraterone acetate PO daily for 4 times, and prednisone PO daily for 3 months. Patients then undergo radical prostatectomy.

ARM III: Patients undergo radical prostatectomy.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate and: Gleason > 8 OR prostatic specific antigen (PSA) > 20 and more than 1 positive core
* Patients with Eastern Cooperative Oncology Group performance scale (ECOG PS) 0 or 1
* Clinical stage T3 or less as demonstrated by abdominal/pelvic computed tomography (CT) or magnetic resonance imaging (MRI) will be selected as the prostate is resectable
* Hemoglobin >= 9.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization
* Platelet count >= 100,000 x 10^9/uL independent of transfusion and/or growth factors within 3 months prior to randomization
* Serum albumin >= 3.0 g/dL
* Glomerular filtration rate (GFR) >= 45 mL/min
* Serum potassium >= 3.5 mmol/L
* Serum total bilirubin =< 1.5 × upper limit of normal (ULN) (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 × ULN, subject may be eligible)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 × ULN
* Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug; must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Clinical stage T4 (invasion into rectum or ureters) significantly increases the morbidity of the surgery

  * Patients with rectal or ureteral invasion will be considered to have unresectable disease
* History of any of the following:

  * Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1year to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign central nervous system [CNS] or meningeal disease which may require treatment with surgery or radiation therapy)
  * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial within 6 months prior to randomization
  * Venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks) within 6 months prior to randomization
  * Clinically significant ventricular arrhythmias within 6 months prior to randomization
* Metastatic prostate cancer
* Baseline moderate or severe hepatic impairment (Child-Pugh class B or C)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Post-surgical potency rate defined as proportion of patients with International Index of Erectile Function score >= 17 | At 12 months
  Each of the experimental arms will be compared to the surgery-only arm, so each test will be a 2.5% level one-sided test to control for the fact that there are two comparisons.

SECONDARY OUTCOMES:
Change in tumor volume on pelvic MRI after neoadjuvant therapy | Baseline to week 13
  Will be correlated with clinical outcomes before and after androgen receptor antagonist ARN-509 or androgen receptor antagonist ARN-509, GnRH agonist, prednisone plus abiraterone acetate.
Number of patients with biochemical recurrence defined using the Prostate Cancer Clinical Trials Working Group 2 definition | Up to 5 years
Number of patients with pathological T0 | Up to 5 years
Number of patients with positive surgical margins | Up to 5 years
Postoperative continence rate as determined by the American Urological Association Symptom Score (AUAss) | Up to 24 months after surgery
Postoperative continence rate as determined by the Sexual Health Inventory for Men | Up to 24 months after surgery
Postoperative continence rate as determined by the Expanded Prostate Cancer Index Composite (EPIC) | Up to 24 months after surgery
Quality of life as assessed by the AUAss questionnaires | Up to 24 months after surgery
Quality of life as assessed by the EPIC questionnaires | Up to 24 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Saum Ghodoussipour, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT02949284/ICF_000.pdf